CLINICAL TRIAL: NCT06501001
Title: Time Restricted Eating and High-Intensity Interval Training to Improve Health in Patients With Metabolic Syndrome
Brief Title: Time Restricted Eating (TRE) and High-Intensity Interval Training (HIIT) to Improve Health in Patients With Metabolic Syndrome (METS)
Acronym: TRE-HIIT-METS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Principal Investigator, Felix Morales Palomo, PhD, University of Castilla-La Mancha
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TRE-HIIT-METS
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Metabolic Syndrome; Exercise; Weight Loss; Obesity; Cardiometabolic Syndrome; Time Restricted Eating
Keywords: Metabolic syndrome; HIIT; Exercise training; Time restricted eating
MeSH Terms: conditions — Metabolic Syndrome; Motor Activity; Weight Loss; Obesity; Intermittent Fasting | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High-Intensity Interval Training (Experimental): High-intensity interval training for sixteen weeks. Three weekly, supervised training sessions.
  Interventions: Behavioral: High-Intensity Interval Training
- Time-Restricted Eating (Experimental): Time-restricted eating for sixteen weeks. Maximal daily eating window of 10 hours
  Interventions: Behavioral: Experimental: Time-Restricted Eating
- High Intensity Interval Training & Time-Restricted Eating (Experimental): High-intensity interval training for sixteen weeks. Three weekly, supervised training sessions.
  Time-restricted eating for sixteen weeks. Maximal daily eating window of 10 hours
  Interventions: Behavioral: High-Intensity Interval Training; Behavioral: Experimental: Time-Restricted Eating
- Control (No Intervention): Information about the recommended level of physical activity for health benefits and a healthy diet will be given.

INTERVENTIONS:
Behavioral: High-Intensity Interval Training — Three weekly, supervised exercise sessions with high intensity. Each session will last for 45 minutes. The intervention period will be sixteen weeks.
  Arms: High Intensity Interval Training & Time-Restricted Eating; High-Intensity Interval Training
Behavioral: Experimental: Time-Restricted Eating — Restricted daily window of caloric intake to a maximum 10 hours. The intervention period will be sixteen weeks.
  Arms: High Intensity Interval Training & Time-Restricted Eating; Time-Restricted Eating

SUMMARY:
Studies in mice provide compelling evidence that feeding/fasting cycles can be altered to produce beneficial effects on weight loss and cardiometabolic health markers in the absence of caloric restriction. Limited research in subjects with metabolic syndrome (MetS) suggests that this feeding paradigm may also apply to human health when combined with an exercise training program, but more research is needed to confirm this hypothesis.

This project will determine the independent and combined effects of high-intensity interval training and time-restricted eating on cardiometabolic factors among overweight or obese patients with MetS.

The intervention period will be sixteen weeks. Before and after the intervention, MetS components (i.e., MetS Z score), body composition, and physical fitness will be measured and compared between groups who are doing either high-intensity interval training, time-restricted eating, both high-intensity interval training and time-restricted eating, or who are in a control group. Physical activity, diet, sleep quality, and intervention adherence will also be measured.

ELIGIBILITY:
Inclusion Criteria:

Metabolic syndrome patients diagnosed according to The International diabetes federation consensus of 2009 (Alberti, et al., Circulation):

* Waist circumference ≥ 92 cm (Men) or ≥ 80 cm (Women).
* Triglycerides ≥ 150 mg/dL (or on drug treatment for elevated triglycerides).
* Reduced HDL-C < 40 mg/dL (Men), < 50 mg/dL (Women) (or on drug treatment for reduced HDL-C).
* Elevated blood pressure, systolic blood pressure ≥ 130 mmHg and/or diastolic blood pressure ≥ 85 mmHg (or treatment with an antihypertensive drug with a history of hypertension).
* Elevated fasting glucose ≥ 100 mg/dL (or drug treatment of elevated blood glucose).
* Age ≥18 to ≤65 years
* Previously inactive (<150 min·wk-1 of the moderate-intensity activity assessed by 7-d IPAQ

Exclusion Criteria:

* Pregnancy, and lactation within 24 weeks of study commencement
* Untreated cardiovascular or renal disease
* Type 1 diabetes
* Any condition associated with exercise intolerance.
* Habitual eating window < 12 hours
* Performing high-intensity training more than once a week
* Body mass variations > 4 kg three months prior to study commencement
* Shift work that includes night shifts

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Metabolic Syndrome Z score | Baseline and after 16 weeks of intervention
  MetS z score will be used to assess the continuous rather than dichotomous (have/not haveMetS) evolution of each MetS component into a compound score. We will calculate the Z score as the difference between the subjects and the threshold value divided by the group standard deviations for each MetS criterion.

SECONDARY OUTCOMES:
Blood lipids profile | Baseline and after 16 weeks of intervention
  Serum concentrations (in mg per dL) of triglycerides, total colesterol, high density lipoprotein after 8-hour fasting
Glycemia | Baseline and after 16 weeks of intervention
  Serum concentrations of glycemia (in mg per dL) after 8-hour fasting
Blood pressure | Baseline and after 16 weeks of intervention
  Systolic and diastolic values of blood pressure measures obtained from the brachial artery after 15 min of supine rest.
Central obesity | Baseline and after 16 weeks of intervention
  Measure waist circumference (cm) in a horizontal plane, midway between the ribs' inferior margin and the iliac crest's superior border.
Body composition | Baseline and after 16 weeks of intervention
  Measurement of the mass of man body compartments (i.e., VAT [visceral adipose tissue] fat mass, fat-free mass, and bone mass) by dual-energy x-ray absorptiometry.
Insulin | Baseline and after 16 weeks of intervention
  Serum concentrations of insulin after 8-hour fasting
Insulin sensitivity | Baseline and after 16 weeks of intervention
  Insulin sensitivity estimated by homeostatic model assessment for insulin resistance (fasting serum insulin concentration (μU/mL) x fasting plasma glucose levels (mmol/L)/22.5)
Cardiorespiratory fitness | Baseline and after 16 weeks of intervention
  Maximum oxygen uptake from a graded exercise test plus a verification test

OTHER OUTCOMES:
Diet intake | Baseline and week 8 of intervention
  Food diary
Daily physical activity | Baseline and week 8 of intervention
  Measurement of daily steps using pedometers
Sleep | Baseline and week 8 of intervention
  Measure by activity monitor
Adherence to high intensity interval training | Week 16
  Number of completed exercise sessions out of those prescribed, in percentage
Compliance to high intensity interval training | Week 16
  Exercise intensity, heart rate in percentage of individual heart rate maximum
Compliance to time-restricted eating | Week 16
  Average daily eating window, in hours
Adherence to time-restricted eating | Week 16
  Average number of days where per week that daily eating window is 10 hours or less.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Castilla La Mancha, Toledo, Spain

IPD SHARING:
Plan to Share IPD: Undecided